CLINICAL TRIAL: NCT05938998
Title: Social Support and Stress Reduction for Caregivers of Young Adults With IDD
Acronym: CareWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Amy Bodde, PhD, MPH, Research Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00149679; 3KL2TR002367-08S1 (NIH)
Record Dates: First submitted 2023-06-29; First posted 2023-07-11 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Burden, Caregiver
Keywords: Caregiver; Down syndrome; Intellectual Disability; Parent; Stress
MeSH Terms: conditions — Caregiver Burden; Down Syndrome; Intellectual Disability | interventions — Yoga; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Support and Yoga (Experimental): This is a single arm trial. This arm includes one hour of a guided social support group and one hour of yoga, weekly for 12 total weeks.
  Interventions: Behavioral: Yoga; Support Group

INTERVENTIONS:
Behavioral: Yoga; Support Group — BEHAVIORAL: Group Exercise Sessions- Yoga. BEHAVIORAL: Social Support Sessions

SUMMARY:
The objective of this study is to evaluate the feasibility and stress reduction impacts of a yoga and support group intervention on caregivers of individuals with intellectual and developmental disabilities.

DETAILED DESCRIPTION:
This is a single arm longitudinal trial. We will recruit up to 40 caregivers of young adults with intellectual and developmental disabilities (IDD). This is a 12-week social support, resources, and stress reduction intervention delivered in person to a group of caregivers of young adults IDD. Participants will be asked to attend one 2 hour group session each week. All sessions will have a 1-hour discussion on resources and social support and 1-hour of yoga. All yoga sessions will be taught by 200 Registered Yoga Teacher certified instructors. Outcome assessments will be collected at baseline and after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* 1) caregiver of a young adult with IDD 2) self-reported ability to participate in a yoga class with no contraindications to participation.

Exclusion Criteria:

* 1) Actively participating in another health lifestyles interventional research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bodde, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From all recruitment methods, 25 caregivers were interested in the intervention and completed the eligibility questionnaire. All 25 were eligible, however the study team was unable to reach 3 participants and 2 more decided not to participate, resulting in a recruitment rate of 80% and an average of 4 participants recruited per month of recruitment. One participant formally dropped out of the study and 3 participants were unavailable for post-test outcomes measurement.
Pre-assignment Details: This was a single-arm pilot trial, therefore all participants were assigned to the intervention arm.
Groups:
- Arm 1: This is a single arm trial, therefore Arm 1 is the intervention arm.
Period: Overall Study
Arm/Group | Arm 1
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of participants
  years | 51.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 2
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants] — Midwestern United States
  Participants
    United States | 20
Family caregiver [Count of Participants; unit: Participants] — Family member versus non-family member caregiver
  Participants | 19

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: We will calculate recruitment rate by dividing the number of participants who enroll by those who were found eligible on the questionnaire.
Time Frame: Baseline
Population: 25 participants completed the eligibility questionnaire. All 25 were eligible, however the study team was unable to reach 3 participants and 2 more decided not to participate, resulting in a recruitment rate of 80%.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 25
Participants | 20

2. Primary Outcome: Session Attendance
Description: The group session leaders will record attendance at weekly sessions. The participants will only be considered present if they complete the entire 2-hour session. The outcome variable will be the number of sessions attended (count) and percentage of attendance out of the total 12 scheduled sessions.
Time Frame: Weeks 1-12 of intervention
Measure: Mean (Standard Deviation); unit: sessions attended
Arm/Group | Arm 1
Number analyzed (Participants) | 19
sessions attended | 8 (3)

3. Primary Outcome: Mean Number of Sessions Attended
Description: Mean number of sessions attended out of 12 possible sessions
Time Frame: From baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Sessions attended
Arm/Group | Arm 1
Number analyzed (Participants) | 19
Sessions attended | 8 (3.5)

4. Primary Outcome: Retention
Description: Calculated as percentage of participants who completed the out of those who enrolled
Time Frame: Weeks 1-12 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 20
Participants | 19

5. Secondary Outcome: Perceived Stress Scale Score
Description: The Perceived Stress Scale will be administered at baseline and post intervention. Individual scores on the Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: 12 weeks
Population: 16 participants were available for outcomes assessment
Measure: Mean (Standard Deviation); unit: Perceived Stress Scale Numeric Score
Arm/Group | Arm 1
Number analyzed (Participants) | 16
Perceived Stress Scale Numeric Score
  Pre-test mean and standard deviation | 22.6 (3.9)
  Post-test mean and standard deviation | 21.3 (4.1)

6. Secondary Outcome: ug/dL Salivary Cortisol
Description: Cortisol will be used of measure physiologic stress collected at baseline and post intervention, self-collected using saliva swabs. Test kits can detect salivary cortisol in the range between 0.012-3.000 ug/dL.
Time Frame: 12 weeks
Population: 13 participants completed saliva samples at both baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Arm 1
Number analyzed (Participants) | 13
ug/dL
  Pre-test mean and standard deviation | 0.63 (0.5)
  Post-test mean and standard deviation | 0.48 (0.2)

7. Secondary Outcome: The Multidimensional Scale of Perceived Social Support (MSPSS)
Description: The Multidimensional Scale of Perceived Social Support (MSPSS) will be given at baseline and post intervention. This measure scores from 12-84 with the higher score indicating more perceived support.
Time Frame: 12 weeks
Population: 15 participants returned surveys.
Measure: Mean (Standard Deviation); unit: MSPSS numeric score
Arm/Group | Arm 1
Number analyzed (Participants) | 15
MSPSS numeric score
  Pre-test mean and standard deviation | 5.1 (1.4)
  Post-test mean and standard deviation | 5.6 (0.8)

8. Secondary Outcome: Modified Caregiver Strain Index
Description: Modified Caregiver Strain Index (MCSI) will be given to participants at baseline and post intervention. Scoring ranges from 26 to 0; a higher score indicates a higher level of caregiver strain.
Time Frame: 12 weeks
Population: 16 participants completed this survey at both baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: Numeric score on MCSI measure
Arm/Group | Arm 1
Number analyzed (Participants) | 16
Numeric score on MCSI measure
  Pre-test mean and standard deviation | 9.2 (5.2)
  Post-test mean and standard deviation | 9.3 (4.1)

9. Secondary Outcome: The Family Empowerment Scale
Description: The Family Empowerment Scale subscales for family and service systems will be administered, at baseline and 12 weeks. Each subscale (family subscale and service subscale) scores from 0-60, with a higher score indicating better family empowerment.
Time Frame: 12 weeks
Population: 16 participants were available for this outcome assessment
Measure: Mean (Standard Deviation); unit: Subscales numeric scores
Arm/Group | Arm 1
Number analyzed (Participants) | 16
Subscales numeric scores
  Family Subscale Pre-test mean and standard deviation | 3.8 (0.6)
  Family Subscale Post-test mean and standard deviation | 4.0 (4.9)
  Services Subscale Pre-test mean and standard deviation | 4.0 (0.6)
  Services Subscale Post-test mean and standard deviation | 4.0 (0.6)

10. Secondary Outcome: The Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index will be administered at baseline and post intervention. Overall scores range from 0 to 21, where lower scores denote a healthier sleep quality.
Time Frame: 12 weeks
Population: 14 participants had valid sleep data at baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: PSQI numeric score
Arm/Group | Arm 1
Number analyzed (Participants) | 14
PSQI numeric score
  Pre-test mean and standard deviation | 7.5 (2.9)
  Post-test mean and standard deviation | 7.6 (4.0)

11. Secondary Outcome: Physical Activity
Description: Moderate to Vigorous Physical Activity and sedentary activity minutes per day assessed by 7 day accelerometer protocol
Time Frame: 12 weeks
Population: Only 11 participants had valid wear time data at both baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Arm 1
Number analyzed (Participants) | 11
minutes/day
  Moderate to Vigorous physical activity Pre-test mean and standard deviation | 31.1 (17)
  Moderate to Vigorous physical activity Post-test mean and standard deviation | 32.6 (21.9)
  Sedentary activity Pre-test mean and standard deviation | 494.1 (95.6)
  Sedentary activity Post-test mean and standard deviation | 487.2 (121.6)

12. Secondary Outcome: Body Mass Index
Description: Body Mass index (body weight in kilograms per height in meters squared) across 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Arm 1
Number analyzed (Participants) | 16
kg/m2
  Pre-test mean and standard deviation | 28.9 (7.4)
  Post-test mean and standard deviation | 28.7 (7.4)

13. Primary Outcome: Acceptability
Description: Number of Participants who Found the Intervention Helpful. Semi-structured interviews were conducted with each caregiver to assess satisfaction with the intervention components.
Time Frame: Between Weeks 12-14
Population: Only 13 of the 20 participants were available for interviews at the end of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Time Frame: From enrollment in the study to the end of measures completion, approximately 14 weeks
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=20)
Pneumonia hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One participant was hospitalized for pneumonia. This was not study related. The participant was discharged and recovered from the illness.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=20)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — One participant reported injuring their back outside of the study. They did not participate in one yoga class but then continued afterward with no problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05938998/Prot_SAP_000.pdf